CLINICAL TRIAL: NCT00005891
Title: Study of Allogeneic Bone Marrow Transplantation Following Cyclophosphamide and Radiotherapy in Patients With Fanconi's Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fairview University Medical Center (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15099; UMN-MT-1982-10; UMN-MT-8210
Record Dates: First submitted 2000-06-02; First posted 2000-06-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-07

CONDITIONS: Fanconi's Anemia
Keywords: Fanconi's Anemia; aplastic anemia; hematologic disorders; rare disease
MeSH Terms: conditions — Fanconi Anemia; Anemia, Aplastic; Hematologic Diseases; Rare Diseases | interventions — Cyclophosphamide

INTERVENTIONS:
Drug: cyclophosphamide
Procedure: Allogeneic Bone Marrow Transplantation

SUMMARY:
OBJECTIVES:

I. Determine the effectiveness of moderate dose cyclophosphamide and total lymphoid radiotherapy in terms of improving the survival and reducing the morbidity following allogeneic bone marrow transplantation in patients with Fanconi's aplastic anemia.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive cyclophosphamide IV over 2 hours on day -6 through -3 and total lymphoid radiotherapy on day -1. Patients undergo allogeneic bone marrow transplantation on day 0.

Patients are followed for at least 100 days.

ELIGIBILITY:
* Diagnosis of severe aplastic anemia with the typical phenotype of Fanconi's anemia: Short stature Hypoplastic radii Skin pigmentation Renal anomalies Chromosomal fragility
* Family history of Fanconi's anemia
* Histocompatible related donor No evidence of excessive in vitro chromosome fragility typical of Fanconi's anemia Normal CBC and bone marrow

Ages: 0 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Weisdorf, Study Chair — Fairview University Medical Center
Locations (1):
- Fairview University Medical Center, Minneapolis, Minnesota, United States